CLINICAL TRIAL: NCT00416897
Title: A Randomised Controlled Trial of Adjunctive Plasma Exchange in Patients With Newly Diagnosed Multiple Myeloma and Acute Renal Failure [MERIT] MyEloma Renal Impairment Trial
Brief Title: Dexamethasone and Chemotherapy With or Without Plasma Exchange in Patients With Newly Diagnosed Multiple Myeloma and Acute Kidney Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000523378; CRUK-MERIT; EU-20670; ISRCTN37161699
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm; Renal Failure
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; renal failure
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Renal Insufficiency | interventions — Drug Therapy; Dexamethasone; Plasmapheresis

INTERVENTIONS:
Drug: chemotherapy
Drug: dexamethasone
Procedure: plasmapheresis

SUMMARY:
RATIONALE: Dexamethasone is used to treat multiple myeloma. Drugs used in chemotherapy may stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Plasma exchange is a process in which certain cells are separated from the plasma in the blood by a machine and then only the cells are returned to the patient. Dexamethasone and plasma exchange may be an effective treatment for acute kidney failure caused by multiple myeloma. It is not yet known whether giving dexamethasone and chemotherapy together with plasma exchange is more effective than giving dexamethasone and chemotherapy alone in treating patients with multiple myeloma and acute kidney failure.

PURPOSE: This randomized phase III trial is studying dexamethasone, chemotherapy, and plasma exchange to see how well they work compared with dexamethasone and chemotherapy alone in treating patients with newly diagnosed multiple myeloma and acute kidney failure.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effect of dexamethasone and cytotoxic chemotherapy with vs without plasma exchange on the likelihood of renal recovery (i.e., dialysis-independent at 100 days) in patients with newly diagnosed multiple myeloma and acute renal failure.

Secondary

* Compare the overall survival of patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Determine the value of renal histology in predicting recovery of renal function in these patients.
* Determine the value of serum free light chain assay in determining disease response and renal function recovery in these patients.

OUTLINE: This is a randomized, controlled, open-label, multicenter study. Patients are stratified according to planned chemotherapy (vincristine and doxorubicin hydrochloride (VA) or VA-like chemotherapy vs thalidomide-containing chemotherapy vs alkylating agent vs other), frequency of chemotherapy courses (1-3 weekly vs 4 weekly), need for dialysis at randomization (yes vs no), and age (< 65 years vs ≥ 65 years). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral dexamethasone, at least twice daily, on days 1-4 and 9-12. Patients undergo plasma exchange by cytocentrifugation or plasmafiltration over 2-3 hours in weeks 1 and 2 (7 treatments total; 4 of them in week 1). Patients then receive planned chemotherapy per local clinician on days 17-100. Chemotherapy may continue after 100 days at the discretion of the local clinician.
* Arm II: Patients receive dexamethasone and planned chemotherapy as in arm I. Quality of life is assessed at baseline, day 100, and 6 and 12 months.

After completion of study treatment, patients are followed at 6 and 12 months and then annually thereafter.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 280 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed multiple myeloma (MM), meeting ≥ 2 of the following criteria:

  * Serum or urine* paraprotein
  * Bone marrow showing > 10% plasma cells
  * Lytic bone lesions NOTE: *The presence of typical myeloma kidney on renal biopsy is considered equivalent to the demonstration of urine paraprotein by electrophoresis
* Acute renal failure attributable to MM, meeting both of the following criteria:

  * Creatinine > 5.65 mg/dL OR urine output < 400 mL/day OR requires dialysis
  * Unresponsive to treatment with fluids and/or treatment of hypercalcemia with bisphosphonates
* No significant intrinsic renal disease unrelated to MM

PATIENT CHARACTERISTICS:

* Platelet count ≥ 50,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* No contraindications to study medication, including the following:

  * Active or recent peptic ulcer
  * Known significant cardiac insufficiency
  * Allergy to study medications
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for MM
* Prior steroid therapy of ≤ 3 days duration for MM allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2003-03; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients alive and dialysis-independent at 100 days

SECONDARY OUTCOMES:
Proportion of patients alive and dialysis-independent at 6 and 12 months
Overall survival
Glomerular filtration rate (calculated or measured) at 15 and 100 days and at 6 and 12 months
Change in serum free light chain levels between days 0 and 15
Response of myeloma to treatment at 100 days and at 6 and 12 months
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Gill Gaskin, MD, Study Chair — Hammersmith Hospitals NHS Trust
Locations (39):
- United Kingdom (39):
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Good Hope Hospital, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Bradford Royal Infirmary, Bradford, England
  - Sussex Cancer Centre at Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St. Helier Hospital, Carshalton, England
  - Saint Richards Hospital, Chichester, England
  - Walsgrave Hospital, Coventry, England
  - Harrogate District Hospital, Harrogate, England
  - Wycombe General Hospital, High Wycombe, England
  - Hull Royal Infirmary, Hull, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester General Hospital, Leicester, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - St. Georges, University of London, London, England
  - Hammersmith Hospital, London, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Nottingham City Hospital, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Hope Hospital, Salford, England
  - Staffordshire General Hospital, Stafford, England
  - Sunderland Royal Hospital, Sunderland, England
  - Royal Cornwall Hospital, Truro, Cornwall, England
  - New Cross Hospital, Wolverhampton, England
  - Cancer Care Centre at York Hospital, York, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Monklands General Hospital, Airdrie, Scotland
  - Dumfries & Galloway Royal Infirmary, Dumfries, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Morriston Hospital NHS Trust, West Glamorgen, Scotland
  - Wrexham Maelor Hospital, Wrexham, Wales